CLINICAL TRIAL: NCT03300245
Title: The Relationship Between the Direction and Degree of Nasal Septal Deviation and Nasal Bone Morphology
Brief Title: Nasal Septum Deviation May Affect Facial Morphologic Parameters.
Acronym: Nasalseptum
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Martina Boshra Shawky, principal investigator, Assiut University
Other Study IDs: 17100286
Record Dates: First submitted 2017-09-27; First posted 2017-10-03 (Actual); Last update posted 2018-07-03 (Actual); Status verified 2018-06

CONDITIONS: Nasal Septal Deviation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with nasal septal deviation: Maxillofacial CT scan
  Interventions: Radiation: Maxillofacial CT

INTERVENTIONS:
Radiation: Maxillofacial CT — clinical and maxillofacial CT data will be tabulated and analysed using by computer software e.g. Statistical Package for the Social Sciences (SPSS)

SUMMARY:
The aim of the study is to evaluate the relationship between the direction and degree of nasal septal deviation with nasal bone morphology , along with factors such as age and gender.

DETAILED DESCRIPTION:
The nasal septum is located in the middle of the nasal cavity and it forms the major part of the nose structure. It is divided into a posterior part by the vomer and perpendicular plate of the ethmoid bone and an anterior part by the quadrangular cartilage .

In the growth period, the nasal septum acts as a growth plate that affects surrounding bones and facial skeletal tissues .Thus, nasal septum deviation affects facial morphologic parameters such as interalveolar distance and maxillary rotation distance, causing compensatory changes in the lateral nasal wall and septal deviation,which are associated with nasal floor and palatal region asymmetries .

Nasal septum deviation is the most common anatomic variation in up to 80% of healthy adults .

From the initial growth stages, the maxillary bone and nasal structure have significant anatomic connections because of their close embryologic development.

The severity of septal deviation also affects the ipsilateral lateral lamina of the cribriform plate width and ipsilateral middle turbinate length . Nasal septal deviation may affect nasal bone growth and facial morphology .Knowledge of nasal morphologic parameters plays an important role in planning successful rhinoplasty and septoplasty operations.

Some morphological characteristics of the nose such as bone length and thickness may present different forms according to factors correlated with age, gender, climate and race.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old who attending to Ear,Nose and throat department out patients complaining of nasal septum deviation causing nasal symptoms are exposed to maxillofacial CT.

Exclusion Criteria:

1. Patients with a history of rhinoplasty,
2. Patients with cranial and facial trauma or bone deformity (e.g. S-shaped septum deviation).
3. Patients with a mass or polyp in the nasal cavity.
4. Patients with adenoid .
5. Patients with nasopharyngeal lesions.
6. Patients with craniofacial anomalies.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: patients attending to E N T clinic
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-08-01 (Estimated); Primary Completion 2019-01-01 (Estimated); Study Completion 2019-03-01 (Estimated)

PRIMARY OUTCOMES:
The nasal deviation angle | 10 minutes
  It will be measured on coronal CT images as the angle between the most deviated point of the septum and the midline which is the line from the crista galli to the palatum
The lateral and intermediate nasal bone thickness | 10 minutes
  The nasal bone thickness will be measured in axial images at the site of the lateral and intermediate osteotomy lines.
  The lateral osteotomy lines run along nasomaxillary suture and intermediate (or midline) osteotomy lines runs along the internasal suture.
  The lateral nasal bone thickness will be measured at the nasomaxillary suture. Intermediate nasal bone thickness was measured at the midpoint between the nasomaxillary suture and the rhinion .
Nasal bone length | 10 minutes
  The nasal bone length will be measured from frontonasal suture to the endpoint of the nasal bone on the sagittal plane
Internasal angle | 10 minutes
  The internasal angle will be measured on coronal CT images at the site of the nasion point

CONTACTS AND LOCATIONS:
Overall Officials: Martina Shawky, Principal Investigator — Assiut University
Locations (1):
- Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hartman C, Holton N, Miller S, Yokley T, Marshall S, Srinivasan S, Southard T. Nasal Septal Deviation and Facial Skeletal Asymmetries. Anat Rec (Hoboken). 2016 Mar;299(3):295-306. doi: 10.1002/ar.23303. Epub 2016 Jan 22. PMID 26677010